CLINICAL TRIAL: NCT05702164
Title: Investigation of Physiotherapy and Rehabilitation Students' Incontinence Knowledge Level and Attitudes Towards Treatment
Brief Title: Physiotherapy and Rehabilitation Students' Incontinence Knowledge Level
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other); Gazi University (Other)
Responsible Party: Principal Investigator, Asli Celik, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2022-1090
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Physiotherapy; rehabilitation; knowledge; incontinence; attitude; therapy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the urinary incontinence knowledge level and attitudes towards treatment in Physiotherapy and Rehabilitation students. With this study, students' knowledge levels about urinary incontinence and treatment parameters will be determined, and it will be possible to show whether there is a difference between genders in terms of knowledge levels.

DETAILED DESCRIPTION:
The aim of the study is to examine the urinary incontinence knowledge level and attitudes towards treatment in Physiotherapy and Rehabilitation students. With this study, students' knowledge levels about urinary incontinence and treatment parameters will be determined, and it will be possible to show whether there is a difference between genders in terms of knowledge levels.

At least 260 students studying in the Physiotherapy and Rehabilitation Department in Turkey will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Physiotherapy and Rehabilitation department in Turkey
* Being volunteer

Exclusion Criteria:

- Failing to complete surveys

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapy and rehabilitation students in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
General information form | Baseline
  Demographic information such as age, gender, height, weight, university will be added to the general information form. In addition, in order to evaluate the level of knowledge of students on urinary incontinence, whether they took courses at the university, whether they followed a patient with urinary incontinence in their internships, the sources they have information about, whether they want to work in this field after graduation, which incontinence assessment methods they know and which treatment methods according to incontinence types, their preferences will be questioned.
Incontinence Quiz | Baseline
  In order to determine the level of incontinence knowledge, Branch et al. It was developed by. The Turkish version study was conducted by Kara et al. made by. The 14-item test is answered as "I agree", "I don't agree" or "I don't know". The correct answer to statements 1, 4, 6, 8, 10, and 11 is "I agree". The correct answer for the remaining statements is "I do not agree". The answer 'I don't know' is calculated incorrectly. The total score ranges from 0 to 14, and a higher score indicates a higher level of knowledge and a more positive attitude towards Urinary Incontinence.
Pelvic Floor Health Knowledge Quiz | Baseline
  The pelvic floor health knowledge quiz investigates the level of pelvic floor health knowledge in the Turkish population and was developed by Al'Deges and Çelenay in 2019. This test consists of 29 questions in three sub-dimensions related to pelvic floor function/dysfunction (8 items), risk and etiology (13 items), diagnosis and treatment (8 items). There is an option of 'Yes' for the positive items used in the test, 'no' for the negative items, and 'I don't know' for the participants who do not have any positive or negative opinion.
Prolapse and Incontinence Knowledge Questionnaire | Baseline
  Prolapse and incontinence information questionnaire Shah et al. It was developed by in 2008 to evaluate incontinence and prolapse knowledge level. Turkish validity and reliability study by Çelenay et al. made by A questionnaire consisting of two 12-item scales; It consists of a urinary incontinence scale to assess women's knowledge of urinary incontinence and a POP scale to assess their knowledge of pelvic organ prolapse. 1 point is awarded for each correct answer and 0 points for each incorrect answer. A score of 0 is given as the answer "I don't know" means lack of knowledge about the current question. Total urinary incontinence and POP scale scores are calculated by summing up the number of correct answers. The total score for each scale can be 0 at the lowest and 12 at the highest.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No